CLINICAL TRIAL: NCT06541028
Title: Reducing Stigma in People Who Inject Drugs With HIV Using a Rapid Start Antiretroviral Therapy Intervention (RS-ART)
Brief Title: Reducing Stigma in People Who Inject Drugs (PWID) With HIV Using a Rapid Start Antiretroviral Therapy Intervention (ART)
Acronym: RS-ART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000035076; 1F32MH138253-01 (NIH); 1R01TW012674-01 (NIH)
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hiv; Drug Use
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PWID in Malaysia- General Population (Experimental): Participants will receive the RS-START strategy (RS-START strategy will be informed and developed in Aims 1 and 2) from prescribing physicians. Participants will complete a survey to assess their experiences with stigma, health behaviors, and other related constructs at baseline, month 1, month 3 and month 6. Data from viral load that are obtained as part of participants' standard of care will be obtained through medical record review.
  Interventions: Behavioral: Rapid-Start ART (RS-ART)
- PWID in Malaysia- Prisoners (Experimental): Participants will receive the RS-START strategy (RS-START strategy will be informed and developed in Aims 1 and 2). Participants will complete a survey to assess their experiences with stigma, health behaviors, and other related constructs at baseline, month 1, month 3 and month 6. Data from viral load that are obtained as part of participants' standard of care will be obtained through medical record review.
  Interventions: Behavioral: Rapid-Start ART (RS-ART)

INTERVENTIONS:
Behavioral: Rapid-Start ART (RS-ART) — ART initiation within 7 days of HIV diagnosis. (RS-ART intervention to be informed and developed in Aims 1 and 2.) RS-ART is a strategy that focuses on clinical decision-making generally based solely on clinical criteria, and later organizing support for mental health, adherence, and management of comorbid conditions only after the patient has initiated ART.

SUMMARY:
This study seeks to develop an RS-ART implementation strategy by utilizing the Delphi method and interviewing experts and PWID regarding their experiences with ART. This strategy will then be pilot tested in a randomized controlled trial (Aim 3). The research will not impact the type of medication and dose prescribed, but rather, how soon providers are able to prescribe ART after diagnosis. The focus of this registration is Aim 3.

DETAILED DESCRIPTION:
Investigators will use a prospective, longitudinal design to pilot test a newly developed RS-ART protocol for PWID with both participants and their HIV clinicians. PWID with HIV will be initiated into the protocol as part of routine care. Aim 3 will be further divided into into aims 3a (general population) and 3b (prisoner population). Aim 3a will not be opened until informed by data collected from Aim 1 and 2. Aim 3b: Will not open until the project is certified by OHRP.

Systematic reviews and cohort studies confirm rapid-start ART (RS-ART) significantly increases ART initiation and viral suppression (VS), central tenets for HIV treatment as prevention (TasP). It focuses on ART initiation within 7 days of diagnosis. Despite recommendations by international agencies and Malaysia's Ministry of Health (MoH) to widely implement RS-ART immediately after diagnosis, it is rarely implemented in Malaysia in key-affected populations (KAPs). Because RS-ART redesigns HIV care by focusing on clinical indicators rather than exploring a patient's worthiness (i.e., stereotypes) for treatment, it has the potential to reduce stigma, though it has not been tested empirically as a stigma reduction strategy in MSM.

Stigma is a well-documented global barrier to health-seeking behavior, engagement in care, and adherence to treatment across a range of health conditions.Stigma emerges when a label associated with a negative stereotype (e.g., MSM, etc.), causing such persons to be seen as separate from and lower in status than others and thus, as legitimate targets of discrimination.

RS-ART, may potentially reduce stigma as a behavioral design intervention (BDI), which can be especially effective where stigma is deeply embedded and difficult to change. BDIs, unlike most extant stigma reduction interventions, use choice architecture, framing and nudging to guide individuals to make specific choices (e.g., immediate ART) or guide behaviors.

ELIGIBILITY:
Inclusion Criteria:

PWID in general population:

* Be a PWID from the general population enrolling into ART services at one of the study's HIV clinics. PWID can include patients injecting opioids, amphetamines, or other combinations of injectable drugs. Some of these patients may be diagnosed with Opioid Use Disorder (OUD).
* Provide informed consent.
* HIV clinicians prescribing ART

  1. Be the HIV clinician who prescribes ART for a PWID in one of the selected clinics.
  2. Be willing to use the RS-ART protocol.
  3. Be at least 18 years old. No minors below age 18 will be enrolled in the study.
  4. Provide informed consent.

PWID in prison population:

* Be a PWID enrolling into ART services at Kajang prison. PWID can include patients injecting opioids, amphetamines, or other combinations of injectable drugs. Some of these patients may be diagnosed with Opioid Use Disorder (OUD).
* Provide informed consent.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
HIV Stigma Framework Scale | Baseline and 6 months
  The scale consists of 24 statements related to the devaluation of people with HIV that are scored on a 5 point Likert-type scale, with higher scores corresponding to higher levels of HIV stigma. Total score range from 24-120. The scale also contains sub-scales for enacted (9 items, score range 9-45), anticipated, (9 items, score range 9-45) and internalized stigma (6 items, score range 6-30).
Substance Use Mechanism Scale | Baseline and 6 months
  All responses are given on a 5-point Likert-type scale, with higher scores indicating greater endorsement of substance use stigma. The scale contains a total of 18 items, with scores ranging from 18-90. Enacted (6 items, score range 6-30), Anticipated (6 items, score range 6-30), and Internalized (6 items, score range 6-30) sub-scales can be created by taking the average of the item responses given for each stigma mechanism respectively.

SECONDARY OUTCOMES:
Viral Load | 6 months
  Mean HIV viral load (in copies/mL) will be obtained through medical record review. A viral load of 200 copies/mL or less is considered 'undetectable' with no risk of HIV transmission.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick L Altice, MD, Principal Investigator — Professor of Medicine (Infectious Diseases) and of Epidemiology (Microbial Diseases)
Locations (3):
- Malaysia (3):
  - Kajang Prison, Kajang
  - Centre of Excellence for Research in AIDS (CERiA) - University of Malaya, Kuala Lumpur
  - Primary Healthcare Centers, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No